CLINICAL TRIAL: NCT06320899
Title: Mid- or High-flex Rods Versus Low-flex Rods of SpineShape System IV for Treatment of Degenerative Lumbar Spine Diseases - a Prospective, Multicenter, Randomized Controlled Non-inferiority Study
Brief Title: Mid- or High-flex Rods Versus Low-flex Rods of SpineShape System IV for Treatment of Degenerative Lumbar Spine Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SpineSave AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SpineShape_CH_001; BASEC 2023-D0092 (Other: Ethics Committee Bern)
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Degenerative Lumbar Spinal Stenosis; Facet Joint Arthrosis; Spondylarthritis; Discopathy; Degenerative Spondylolisthesis; Instability Lumbar Spine
MeSH Terms: conditions — Spondylarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SpineShape System IV straight rod elastic (Experimental): Dynamic stabilization of lumbar segments using SpineShape System IV straight rod elastic (high-flex)
  Interventions: Device: SpineShape System IV straight rod elastic
- SpineShape System IV straight rod medium (Experimental): Dynamic stabilization of lumbar segments using SpineShape System IV straight rod medium (mid-flex)
  Interventions: Device: SpineShape System IV straight rod medium
- SpineShape System IV straight rod stiff (Active Comparator): Dynamic stabilization of lumbar segments using SpineShape System IV straight rod stiff (low-flex)
  Interventions: Device: SpineShape System IV straight rod stiff

INTERVENTIONS:
Device: SpineShape System IV straight rod elastic — Implantation of SpineShape System IV straight rod elastic
  Arms: SpineShape System IV straight rod elastic
Device: SpineShape System IV straight rod medium — Implantation of SpineShape System IV straight rod medium (mid-flex)
  Arms: SpineShape System IV straight rod medium
Device: SpineShape System IV straight rod stiff — Implantation of SpineShape System IV straight rod stiff (low-flex)
  Arms: SpineShape System IV straight rod stiff

SUMMARY:
The purpose of this multi-center, randomized, clinical study is to show that the treatment of degenerative lumbar spine with high- or mid-flex rods is not inferior to the treatment with low-flex rods in terms of clinical and safety-related results.

The primary aim is to compare the reduction in back pain after the treatment with high- or mid-flex rods with that after treatment with low-flex rods. Secondary, the functionality after treatment with high- or mid-flex rods will be compared to that after treatment with low-flex rods.

DETAILED DESCRIPTION:
Dynamic stabilization systems for the lumbar spine are no novelty. The SpineShape System IV builds on the experience of previous systems and attempts to provide additional benefits primarily through three different and relatively elastic rod stiffnesses. 126 subjects with degenerative symptoms in 1 to 2 segments of the lumbar spine L1 to S1 will be recruited. The participants will be randomized in a 1:1:1 ratio to undergo implantation of either the elastic (experimental product group 1), medium (experimental product group 2) or stiff rod (comparison product group).

The aim of the study is to show that the treatment of degenerative lumbar spine with elastic or medium rod variants is not inferior to treatment with hard rods in terms of clinical and safety-related results. This is checked by completing a questionnaire before the surgical procedure and 3 months, 12 months, 24 months and 60 months after the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* degenerative symptoms in 1 to 2 segments in the lumbar spine L1-S1
* signed informed consent of participant
* confirmation of the participant that the attendance of follow-up visits are intended
* Body-Mass-Index < 32
* Pedicle screw axis distance < 30mm
* one or more of the following indications:

  * (dynamic) stenosis in the spinal canal
  * neuroforaminal stenosis
  * facet joint syndrome / spondylarthrosis
  * discopathy (recurrent disc hernia)
  * degenerative spondylolisthesis (Meyerding <1)
  * instability (hypermobility with antelishtesis, hypomobility with retrolisthesis if decompressed)

Exclusion Criteria:

* missing bone structure, e.g. due to congenital anomalies or sever anatomical deformities that make anchoring of the implant impossible
* damaged structural tissue, e.g. due to a bone fracture
* application to the thoracic or cervical spine
* pronounced idiopathic scoliosis
* spondylolisthesis > Meyerding grad 1
* isthmic spondolylysis
* bone tumor
* osteochondrosis modic type I, II or III
* osteoporosis, which could impair screw anchoring
* history with third party implants
* patients with an active local or systemic infection
* known allergy to titatnium alloys
* skeleton in growth (epiphyseal joints not closed)
* severe muscular neuronal or vascular disease
* immunosuppresive therapy
* long-term therapy with cortisone
* heavy smokers (regular consumption of more than six cigarettes per day), drug addicts and alcoholics
* chronic pain patients
* incapable of judgment or emergency situation
* implantation during pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2031-08-31 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) lower back pain | 24 months post-implantation
  self reported back pain intensity using Visual Analogue Scale system. 0 "no pain" to 10 "worst possible pain"

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) leg pain | 3, 12, 24, 60 months post-implantation
  self reported leg pain intensity using Visual Analogue Scale system. 0 "no pain" to 10 "worst possible pain"
walking duration | 3, 12, 24, 60 months post-implantation
  self reported walking duration in 5 categories (0-5 min, 6-15 min, 16-30 min, 31-60 min and >60min)
medication consumption | 3, 12, 24, 60 months post-implantation
  use of none, mild pain medication, non-steroidal anti-inflammatory drugs, opioids, and/or antidepressiva documented in patient's health records
adverse events | after 3, 12, 24, 60 months post-implantation
  adverse events related to the device (e.g. screw loosening, screw breakage, torn rod, slipped rod or too short rod)
segmental mobility index level | 3, 12, 24, 60 months post-implantation
  measuring the segmental mobility at index level to verify the preservation of the mobility. an average mobility per segment of >1° is considered a success
ability to work/ activity (for retirees) | 3, 12, 24, 60 months post-implantation
  self reported ability to work or activity (for retirees) in 5 categories (0%, 25%, 50%, 75%, 100%)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Cathrein, Dr.med., Principal Investigator — Hirslanden Klinik Linde
Locations (2):
- Switzerland (2):
  - Spital Aarberg, Aarberg
  - Hirslanden Klinik Linde, Biel